CLINICAL TRIAL: NCT05062551
Title: Effectiveness of Three Steps Hysteroscopic Repair of Post Caesarean Isthmocele in Patients With Post Menstrual Spotting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mervit Sersy (Other)
Responsible Party: Sponsor-Investigator, Mervit Sersy, Assistant professor, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0305227
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Intervention Model Description: the 50 patients will be subjected to three steps hysteroscopic resection of an isthmocele by removing the distal edge of the niche then the proximal edge and lastly ball cauterization of the floor of the pouch of the isthmocele. Post-operative trans vaginal ultrasound and follow up for 2 menstrual cycles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervetion group (Experimental): 50 patients complained of post-menstrual bleeding with confirmed presence of isthmocele. After written consent, the patient will be subjected to three steps hysteroscopic resection of an isthmocele by removing the distal edge of the niche then the proximal edge and lastly ball cauterization of the floor of the pouch of the isthmocele. Post-operative trans vaginal ultrasound and follow up for 2 menstrual cycles.
  Interventions: Procedure: three steps hysteroscopic resection of an isthmocele

INTERVENTIONS:
Procedure: three steps hysteroscopic resection of an isthmocele — removing the distal edge of the niche then the proximal edge and lastly ball cauterization of the floor of the pouch of the isthmocele. Post-operative trans vaginal ultrasound and follow up for 2 menstrual cycles.

SUMMARY:
Isthmocele is one complications of repeat cesarean sections which is considered as a pocket .that accumulate menstrual blood causing post- menstrual spotting Hysteroscopic resection of the edges of the isthmocele is considered the best treatment option available up to date. Aim of the work: Asses the effectiveness of three steps method resection using hysteroscopy of an isthmocele in patients complained of post -menstrual bleeding with confirmed presence of isthmocele.

.

DETAILED DESCRIPTION:
The incidence rate of cesarean deliveries has been dramatically increased in Egypt.(1) Isthmocele is one of the known complications of repeat cesarean sections.(2) Post- menstrual spotting and many other gynecological complains have been correlated to this isthmocele which is considered as a pocket that accumulate menstrual blood. (3) Hysteroscopic resection of the edges of the isthmocele is considered the best treatment option available up to date.(4) Aim of the work: Asses the effectiveness of three steps method resection using hysteroscopy of an isthmocele in patients complained of post-menstrual bleeding with confirmed presence of isthmocele.

Patients: 50 patients complained of post-menstrual bleeding with confirmed presence of isthmocele. After written consent, the patient will be subjected to three steps hysteroscopic resection of an isthmocele by removing the distal edge of the niche then the proximal edge and lastly ball cauterization of the floor of the pouch of the isthmocele. Post-operative trans-vaginal ultrasound and follow up for 2 menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* female
* previous cesarean sections
* complain post menstrual spotting

Exclusion Criteria:

* other genital tract abnormality
* other uterine causes pf bleeding residual myometrial thickness less than 3mm

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
size of the the niche post operatively | 2 months
  effectiveness of three steps method resection using hysteroscopy of an isthmocele

SECONDARY OUTCOMES:
improving of post menstrual bleeding | 2months
  no more post menstrual spotting

CONTACTS AND LOCATIONS:
Overall Officials: Mervat MD Elsersy, MD, Principal Investigator — Assistant professor
Locations (1):
- Shatby Maternity University Hospital, Alexandria, El-Khartoum Square, Egypt